CLINICAL TRIAL: NCT03230942
Title: Effect of Pre-operative Patient Education Program on Functional Outcomes After Total Knee Arthroplasty
Brief Title: Effect of Pre-op Patient Education on Functional Outcomes After TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Gilmar Moraes Santos, PhD, University of the State of Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UDESantaCatarina
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Knee Arthropathy
Keywords: patient education; arthritis; knee; arthroplasty; gait
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All patients will be assessed for functional outcomes by a rater blinded to the study arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient education program (Experimental): Pre-operative education and pos-operative rehabilitation in individuals will be undergo knee arthroplasty.
  Interventions: Other: Pre-operative education; Other: Pos-operative rehabilitation
- Control - only pos-op rehabilitation (Active Comparator): Pos-operative rehabilitation in individuals will be undergo knee arthroplasty.
  Interventions: Other: Pos-operative rehabilitation

INTERVENTIONS:
Other: Pre-operative education — Verbal and booklet about symptoms and physical conditions pos knee replacement
  Other Names: Patient education program
  Arms: Patient education program
Other: Pos-operative rehabilitation — Physical therapy treatment

SUMMARY:
This study aims to evaluate the effect of preoperative patient education program on functional mobility, gait, postural control, and kinesiophobia level in subjects with TKA. Patients of both gender will be recruited unilaterally in the city of Florianopolis and referred by an orthopedist to the Physiotherapy Clinic of UDESC. They are divided into two groups: one that will receive verbal guidance and a booklet with related information such as your physical condition as well as signs and symptoms in the postoperative period and a group that will receive only verbal guidance.Both groups will be evaluated by a blind evaluator in the preoperative and postoperative periods (6 weeks and 6 months). The evaluations will be divided into five stages. Anthropometric measurements of the individual will be made and then the WOMAC functionality questionnaire and the Kinesiophobia Cover Scale will be applied.Then the individual will walk for 5 meters for three-dimensional gait analysis and electromyographic analysis of the quadriceps and femoral biceps. The evaluation of functional mobility by Timed Up And Go and assessment of postural control in an equilibrium platform will also be performed. Statistical data will be analyzed by analysis of variance 3x2 considering factor time (pre, post 6 weeks and post 6 months) and groups (with and without information leaflet). The value of p will be 0.05.

DETAILED DESCRIPTION:
The study will be developed in the dependencies of the Laboratory of Biomechanics of the Center for Health Sciences and Sports of UDESC. In the preoperative period the subjects will be informed about their physical conditions as well as signs and symptoms of the postoperative period. One group (GI) will receive this information verbally and one leaflet while the other group (GC) will receive only verbal information. The allocation in these groups will be through a lottery, carried out by a member of the team who will not participate in the evaluation stages.

This staff member will read the booklet individually for each GI participant, in a reserved room, before handing out the leaflet to take home. GI participants will be encouraged to reread the information in the home environment and will be asked about the completion of this in the following steps by the staff member responsible for the blinding.

All participants included in the study will perform the kinematic, kinetic and electromyographic gait analysis as well as evaluation of fear of movement, functional mobility and self-perceived functionality in the pre (baseline)-and postoperative period (6 weeks and after 6 months).

The total duration of each evaluation will be approximately 2 (two) hours and 30 (thirty) minutes and all collections will be carried out by the same team. The participant will be allowed to stop the test if they feel pain or become fatigued.

ELIGIBILITY:
Inclusion Criteria:

* Literate;
* Elective submission of unilateral total knee arthroplasty (TKA) due to osteoarthrosis
* Individuals without other arthroplasties in the lower limb in the last 6 months;
* Range of motion greater than 90 degrees or operated contralateral knee.

Exclusion Criteria:

* Associated condition that impedes performance in gait tests, including significant osteoarthrosis in the contralateral knee or hips (defined as pain greater than or equal to 5 on the analog visual pain scale);
* Absence or abandonment in the study follow-up sessions.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Timed up And Go Test score | pre-operative; 6 weeks; 6 months
  The timed up and go requires a patient to rise from a chair walk three meters around a piece of tape and return to the chair again as quickly as possible. The TUG has good inter-rater and intra-rater reliability and validity for functional testing in older adults at risk for falls. The test is easy to administer and can be completed in two to three minutes.Change from baseline (pre-operative) in the functional mobility. The variable will be measured in seconds.

SECONDARY OUTCOMES:
EMG activity | pre-operative; 6 weeks; 6 months
  Electromyographic activity of rectus femoris, vastus lateralis, vastus medialis, vastus medial and gastrocnemius by NORAXON WIRELESS EMG. Change from baseline (pre-operative).The variable will be measured in % of maximal voluntary contraction.
Kinematics | pre-operative; 6 weeks; 6 months
  Gait analysis by VICON three-dimensional ,10-camera motion capture system.The outcome measurement is assessed at pre-operation, six weeks and six month after operation. Change from baseline (pre-operative). The variable will be measured in degrees.
Kinetics | pre-operative; 6 weeks; 6 months
  Gait analysis by AMTI plate force. The outcome measurement is assessed at pre-operation, six weeks and six month after operation. Change from baseline (pre-operative). The variable will be measured in newtons

OTHER OUTCOMES:
kinesiophobia | pre-operative; 6 weeks; 6 months
  Fear of movement. The variable will be measured in points (score).

CONTACTS AND LOCATIONS:
Overall Officials: Gilmar M Santos, PhD, Principal Investigator — University of State of Santa Catarina
Locations (1):
- Center for Health and Sport Sciences, Florianópolis, Santa Catarina, Brazil

DOCUMENTS (3):
  • Informed Consent Form (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT03230942/ICF_000.pdf
  • Statistical Analysis Plan (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT03230942/SAP_001.pdf
  • Study Protocol (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT03230942/Prot_002.pdf